CLINICAL TRIAL: NCT01440842
Title: An Open-label, Single-centre, Randomised Controlled Trial to Assess the Safety and Efficacy of Automated Closed-loop Blood Glucose Control in Comparison With Standard Care in Adults in Intensive Care Unit
Brief Title: Closed Loop Glucose Control in Intensive Care Unit
Acronym: CLASSIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: European Commission (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Lalantha Leelarathna, Clinical Research Associate, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLASSIC 01
Record Dates: First submitted 2011-09-22; First posted 2011-09-27 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Stress Hyperglycaemia
Keywords: Stress hyperglycaemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-loop (Model Predictive Control Algorithm) (Experimental)
  Interventions: Other: Closed-loop insulin delivery
- Open loop (Standard treatment) (Active Comparator)
  Interventions: Other: Standard IV insulin infusion sliding scale

INTERVENTIONS:
Other: Closed-loop insulin delivery — Intravenous infusion delivery of Actrapid insulin and dextrose, dose calculated by Model Predictive Control (MPC) algorithm, based on continuous glucose sensor readings.
  Arms: Closed-loop (Model Predictive Control Algorithm)
Other: Standard IV insulin infusion sliding scale — Standard intravenous insulin infusion sliding scale as per intensive care unit protocol.
  Arms: Open loop (Standard treatment)

SUMMARY:
The purpose of this study is to assess the efficacy, safety and feasibility of a computer-based control algorithm to control glucose levels in adults in intensive care unit, in comparison to standard care.

DETAILED DESCRIPTION:
This will be a single centre, open-label, randomised, parallel design, feasibility study conducted at Neurosciences Critical Care Unit (NCCU), Addenbrooke's hospital, Cambridge, UK. Study will aim for 24 adult subjects (12 participants in each arm of the trial) and study will last for up to 49 hours in each subject. Subjects will have a commercially available Conformité Européenne(CE) marked subcutaneous glucose sensor inserted at the start of the study. Glucose data from the sensor will be transmitted to a small bedside tablet computer, containing the algorithm which will determine insulin infusion rates aimed at maintaining glucose level between 6.0 - 8.0 mmol/L. The advice from the algorithm will be sent to the infusion pump via USB cable and insulin will be delivered intravenously. The system will also deliver intravenous glucose via a second infusion pump at times of low glucose levels. Samples for reference glucose values will be obtained either from an arterial line or central venous cannula and will be analysed using standard blood gas analyser in real time. Subjects randomised to standard care will receive intravenous insulin based on current treatment guidelines at the Neurosciences critical care unit (NCCU), Addenbrooke's Hospital, Cambridge, UK.

The primary outcome is time spent in target glucose range between 6.0 to 8.0 mmol/L as recorded by reference glucose. Secondary outcomes are the time spent with glucose levels above and below target, as recorded by reference glucose, and sensor accuracy. Safety includes evaluation of significant hypoglycaemia and hyperglycaemia and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Admitted to Neurosciences critical care unit; (all patients are eligible regardless of admitting diagnosis except where specified under exclusion criteria)
* Stay in intensive care unit expected to be at least 48 hours
* At least one of the following conditions applies:
* Not on insulin infusion and single confirmed reference blood glucose level > 10.0 mmol/l
* Already on insulin infusion including those subjects with pre-existing diabetes.

Exclusion Criteria:

* Patients with diabetic ketoacidosis or hyperosmolar hyperglycaemic non-ketotic coma (HONK)
* Patients who are receiving therapeutic hypothermia
* Known or suspected allergy to insulin
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient (i.e. liver failure, other fatal organ failures)
* Patients with significant abnormalities of blood clotting.
* Moribund patients likely to die within 48 hours
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose values in target range (6.0 - 8.0 mmol/l) as recorded by reference glucose measurements. | Up to 49 hours in each subject.
  Definition of Reference glucose = Blood Glucose level measured by arterial blood gas analyzer.
  During the study subjects will have the reference glucose measured every 1 hour and this is used for the calculation percentage glucose values.

SECONDARY OUTCOMES:
Percentage of glucose values in range (4.0 - 10.0 mmol/l) as recorded by reference glucose measurements. | Up to 49 hours in each subject
  Definition of Reference glucose = Blood Glucose level measured by arterial blood gas analyzer.
  During the study subjects will have the reference glucose measured every 1 hour and this is used for the calculation percentage glucose values.
Percentage of glucose values <4.0 mmol/l and >8.0 mmol/l as recorded by reference glucose measurements. | Up to 49 hours in each subject.
  Definition of Reference glucose = Blood Glucose level measured by arterial blood gas analyzer.
  During the study subjects will have the reference glucose measured every 1 hour and this is used for the calculation percentage glucose values.
Percentage of glucose values > 10.0 mmol/l as recorded by reference glucose measurements. | Up to 49 hours in each subject,
  Definition of Reference glucose = Blood Glucose level measured by arterial blood gas analyzer.
  During the study subjects will have the reference glucose measured every 1 hour and this is used for the calculation percentage glucose values.
Mean and standard deviation of reference glucose measured using arterial blood gas analyzer | Up to 49 hours in each subject.
  Definition of Reference glucose = Blood Glucose level measured by arterial blood gas analyzer. This is reported in mmol/L
  During the study subjects will have the reference glucose measured every 1 hour and this is used for the calculation of mean (mmol/L) and standard deviation which will reflect the efficasy of closed loop insulin delivery.
Mean and median absolute and relative difference between matched pairs of subcutaneous glucose sensor and reference plasma glucose. | Up to 49 hours in each subject.
  For a given subcutaneous glucose sensor value, difference between the sensor and the reference glucose will be calculated. Example - Reference glucose 10 mmol/L and sensor glucose 12 mmol/L, therefore absolute difference will be 2 mmol/L. Mean and median of these deviations will be reported in mmol/L. The term relative implies that data has been converted to a percentage deviation from reference glucose.
Time to reach target glucose | Up to 49 hours in each subject.
Insulin infusion rates | Up to 49 hours in each subject.
Frequency and magnitude of significant hypoglycaemic (< 3.0 mmol/L), severe hypoglycaemic (<2.0 mmol/L) and significant hyperglycaemic (> 15mmol/l) episodes. | Up to 49 hours in each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, BSc MSc PhD, Principal Investigator — University of Cambridge; Rowan Burnstein, MBBS FRCA PhD, Principal Investigator — Addenbrooke's Hospital, Cambridge, United Kingdom
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Leelarathna L, English SW, Thabit H, Caldwell K, Allen JM, Kumareswaran K, Wilinska ME, Nodale M, Mangat J, Evans ML, Burnstein R, Hovorka R. Feasibility of fully automated closed-loop glucose control using continuous subcutaneous glucose measurements in critical illness: a randomized controlled trial. Crit Care. 2013 Jul 24;17(4):R159. doi: 10.1186/cc12838. PMID 23883613